CLINICAL TRIAL: NCT03994458
Title: The Efficacy and Compliance of Using A Smartphone Application in Treating Non-Specific Low Back Pain Among Office Employees: A Randomized Controlled Trial
Brief Title: The Efficacy of A Smartphone Application in Treating Non-Specific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Khader Almhdawi, Associate professor, Jordan University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20180429
Record Dates: First submitted 2019-06-17; First posted 2019-06-21 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Low Back Pain
Keywords: Musculoskeletal Rehabilitation; Smartphone application; Occupational Stress
MeSH Terms: conditions — Low Back Pain; Occupational Stress

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial, double blinded
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinded evaluators and participants are not aware which version of the program they got.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Participants get the full program for 6 weeks.
  Interventions: Behavioral: Smartphone Full version application
- Placebo (Placebo Comparator): Participants get the placebo program for 6 weeks.
  Interventions: Behavioral: Samartphone limited version application

INTERVENTIONS:
Behavioral: Smartphone Full version application — Android smartphone experimental application include: rehabilitative self-administered evidence-based exercises (Strengthening and stretching), ergonomics, and education related to low back pain. The application includes videos, photos, text, and reminders.
  Other Names: Experimental
  Arms: Experimental
Behavioral: Samartphone limited version application — Android smartphone placebo application include: ineffective content that does not help in treating low back pain. The application includes only five posts in the general instruction and advises section about proper nutrition and few irrelevant reminders.
  Other Names: Placebo control
  Arms: Placebo

SUMMARY:
Evaluating the efficacy of a newly developed self-monitored mobile application in reducing office workers low back pain.

DETAILED DESCRIPTION:
II. Introduction and Hypothesis of the Study:

Around 12% to 33% of the adult workforce are affected by low back pain (LBP) each year. Furthermore 70% to 95% of the adults are predicted to have back pain at least once in their lifetime (Van Tulder et al., 2006, Karthikeyan et al., 2013). There are numerus applications for self-management of LBP. These applications provided patients with cost-effective alternative management for their LBP. However, most of these available applications are of a low quality, because they were developed without an evidence-based vision (Machado et al., 2016).

Hypothesis:

1. All participants who will use the full access of the LBP application for six weeks will demonstrate significant decrease in low back pain intensity as measured by Visual Analogue Scale (VAS).
2. All participants who will use the full access of the LBP application for six weeks will demonstrate significant decrease in disability as measured by Oswestry Disability Index (ODI).
3. All participants who will use the full access of the LBP application for six weeks will demonstrate significant perceptual satisfaction and gained benefit as measured by self-rated survey questions.

III. Aims of the study: This study aims to evaluate the efficacy and compliance in using a standardized evidence-based LBP application among office employees who suffer from non-specific LBP, in randomized controlled trial.

IV. Materials and Methods: A smartphone application will be programed to deliver home-based exercises and advices targeting LBPP. 30 participants who has LBP, had been at least 5 years office worker have a 5 hours of working, will be recruited for a randomized controlled trial, participants who have any spine or spinal cord disease will be excluded. Participants will be compared according who will get full access to the application for non-specific LBP management with those who will get a limited version of the application. Both groups will use their versions of the application for 6 weeks, a follow-up will be done after 6 weeks. Visual Analog Scale (VAS), will be used to assess intensity of the LBP, and Oswestry Disability Index (ODI) will be used to assess the disability that had been caused by LBP. Descriptive statistics will be represented in means and standard deviations. Change scores between groups (experimental vs control) will be compared using ANCOVA model.

ELIGIBILITY:
Inclusion Criteria:

1. Being office worker for at least 5 years with at least 5 hours of working daily behind the desk.
2. Middle age adults, age between 30 and 55 years old.
3. Complains of LBP at least for 3 months measured by self-report
4. Scored at least 3 point on a 0-10 Visual Analog Scale.
5. Owning an android smartphone.

Exclusion Criteria:

1. Pregnancy.
2. Diagnosed with disc herniation with radiculopathy pain.
3. Structural deformities as in Scoliosis, or Kyphosis, or Lordosis.
4. Spinal tumor.
5. Ankylosing spondylitis, spondylolisthesis.
6. Had a spine surgery or significant trauma in the past 6 months.
7. Low mental ability of not being able to use smartphone.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Change in Visual Analog Scale (VAS) scores | Change from basleine to 6 weeks will be assessed.
  A measure used to evaluate pain related to low back pain. Score range is 0-10, where higher scores indicate more pain.
Change in Oswestry Disability Questionnaire (ODQ) scores | Change from basleine to 6 weeks will be assessed.
  A measure used to evaluate disability related to low back pain. Score range is 0-100, where higher scores indicate more disability.

SECONDARY OUTCOMES:
Change in 12-item Short Form Health Survey (SF-12) scores | Change from basleine to 6 weeks will be assessed.
  A measure of health related quality of life includes Physical Component Summary (PCS) and Mental Component Summary (MCS) scores. Score range is 0-100, where higher scores indicate better health related quality of life.
Change in Depression, Anxiety, and Stress Scale (DASS21) scores | Change from basleine to 6 weeks will be assessed.
  A measure used to assess mental health symptoms over the last week. Score range is 0-21, where higher scores indicate worse mental health.
Change in Pittsburgh Sleep Quality Index (PSQI) scores | Change from basleine to 6 weeks will be assessed.
  The PSQI assess sleep quality over previous month.Score range is 0-21, where higher scores indicate worse sleep quality.
Change in International Physical Activity Questionnaire -short form (IPAQ-SF) scores | Change from basleine to 6 weeks will be assessed.
  A measure collects the occurrence and time of physical activity with continuous high, moderate and low intensity for at least ten minutes during the previous 7 days. A higher score in this measure indicates higher physical activity level.

CONTACTS AND LOCATIONS:
Overall Officials: Khader Almhdawi, Ph.D, Principal Investigator — Jordan University of Science and Technology
Locations (1):
- Jordan University of Science and Technology, Irbid, Jordan